CLINICAL TRIAL: NCT01217775
Title: A Phase 3 Study of the Use of PH80 for Acute Management of the Symptoms of Premenstrual Dysphoric Disorder
Brief Title: Intranasal PH80 Spray for Acute Management of the Symptoms of Premenstrual Dysphoric Disorder
Acronym: PH80-PMD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pherin Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PH80 CL019
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Premenstrual Dysphoric Disorder
Keywords: PMDD, Premenstrual, Dysphoria, Mood Swings, Bloating.
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PH80 intranasal spray (Experimental): Start using study medication on 14th of the cycle, or the day symptoms start to bother, or if no symptoms on day 21st of the cycle but no later than day 21st of the cycle, up to 6-times per day, and continuing until day 2-3 of the menses
  Interventions: Drug: PH80
- Placebo intranasal spray (Placebo Comparator): Start using study medication on 14th of the cycle, or the day symptoms start to bother, or if no symptoms on day 21st of the cycle but no later than day 21st of the cycle, up to 6-times per day, and continuing until day 2-3 of the menses
  Interventions: Drug: Placebo intranasal spray

INTERVENTIONS:
Drug: PH80 — PH80 intranasal spray 800 nanograms
  Arms: PH80 intranasal spray
Drug: Placebo intranasal spray — Placebo intranasal spray
  Arms: Placebo intranasal spray

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety in double-blind, randomized, placebo-controlled clinical trials of self administered PH80 intranasal spray for the acute management of cycle related symptoms in women who regularly experience premenstrual dysphoric disorder (PMDD).

DETAILED DESCRIPTION:
Premenstrual disorders are characterized by negative mood, behavioral, and physical symptoms that occur consistently for several days to two weeks before menses, that can disrupt normal functioning, and that subside during the postmenstrual phase of the cycle. Marked irritability, marked depressed mood, marked anxiety, overeating of specific food cravings, mood swings, lack of energy, and pain are among the most common symptoms of moderate to severe premenstrual disorders.

It is estimated that 75% women of reproductive age (menarche to perimenopause) experience physical and behavioral symptoms premenstrually and in 40% women symptoms are intense (moderate to severe) and require medical attention. For 3-8 % women premenstrual symptoms are severe enough to interfere with work and interpersonal relationships. Premenstrual Dysphoric Disorder (PMDD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) research criteria, represents the more severe and disabling end of the premenstrual disorders spectrum. For women with severe premenstrual symptoms or PMDD, these symptoms are bothersome enough to produce an impact on psychological and/or occupational functioning, and professional attention is required.

Selective serotonin reuptake inhibitors (SSRIs) fluoxetine, sertaline and paroxetine have been approved by the United States Food and Drug Administration (FDA) as a chronic treatment for PMDD, however the use of SSRIs significantly increases the risk of suicide in adolescents and young adults. Antidepressants are also associated with significant relapse during short and long term treatment of PMDD. Contraceptives are also prescribed to treat moderate and severe premenstrual symptoms, but besides the severe adverse effects (drospirenone and ethinyl estradiol) they re not the treatment choice for women willing to become pregnant.

Pherin Pharmaceuticals synthesized a number of pherines and screened them for biologic activity in vitro. PH80 is a pherine shown to bind to a subset of peripheral receptors in nasal chemosensory neurons. Pherines such as PH80 are thought to exert their activity by rapid stimulation of the hypothalamus, which does not require systemic uptake and distribution. PH80 is being investigated as a potential treatment in women that suffer the cycle related symptoms of Premenstrual Dysphoric Disorder.

Each single administration of PH80 to be tested in this study will deliver a similar amount of PH80 (800 nanogram) to the nasal passages as was found in previous investigations (Pherin Clinical Study #PH80 CL003, #PH80 CL015 and #PH80 CL016) to improve premenstrual symptoms in PMDD patients when administered intranasally on an acute basis.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 to 43 years, with regular menstrual cycles between 22 - 35 days in length inclusive.
* Women of childbearing potential may participate if they are not pregnant or breast feeding, and if they agree to use one of the following methods of contraception throughout the study: abstinence, intrauterine device, condom and foam, diaphragm and spermicide, vasectomy and spermicide, tubal ligation and spermicide, oral contraceptives and barrier method. Women using oral contraceptives must have been on a stable dosing regimen for at least 6 months prior to study entry and must agree to continue on that same dosing regimen throughout all phases of the study.
* Patients who reported at least a 1-year history of regularly experiencing PMDD.
* Patients who are able to read and understand the Informed Consent document; are willing and able to comply with the protocol; and who had read, understood, and voluntarily signed the written Informed Consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* Patients who fail to meet the study criteria for PMDD
* Patients with active diabetes mellitus, neurological, cardiac, renal, hepatic, or pulmonary disease, or with any other significant medical or gynecological abnormality or condition, as determined by physical examinations and/or clinical laboratory tests.
* Patients diagnosed with Major Depressive Disorder or Bipolar Depression.
* Patients with an acute or chronic condition that at the judgment of the clinical Investigator could harm the patient and/or alter the outcome of the study. Additional clinical examinations and symptom assessment will be performed at this time to determine continuing eligibility for study participation.
* Patients who used any intranasal medication other than study drug within 14 days prior to study entry and/or during the Run-In and/or Treatment Phases of the study.
* Patients with other clinical conditions or diseases, or those who were taking concomitant medications, which in the clinical judgment of the Investigator could place the patient at undue risk, interfere with study participation, or confound the results of the study.
* Patients with current or last 2 years history of substance abuse.
* Patients who had a positive urine drug screen for any of the following: amphetamines, barbiturates, cocaine metabolites, opiates, benzodiazepines, and/or cannabinoids.
* Patients who had been treated previously with PH80.
* Patients who had participated in another research study or received another investigational drug within 30 days prior to study entry or during the study.
* Patients who used any other exclusionary prescription and/or nonprescription medications as specified in the study protocol (described in this report) within 14 days prior to study entry and/or during the Run-In and/or Treatment Phases of the study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1400 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Daily Record of Severity of Problems (DRSP)scores | Daily DRSP sores
  Primary outcome meassure: difference between average luteal phase DRSP total scores from 2 qualification cycles and average luteal phase DRSP socores from 6 treatment cycles.

SECONDARY OUTCOMES:
Patient Global Evaluation (PGE) | Daily PGE scores
  Secondary outcome measures include: each of the 11 individual items of the DRSP, scheduled patient and Investigator global evaluations of the patients' PMDD symptoms, including patient-rated Global Evaluations (PGE) and Investigator rated Clinical Global Impression (CGI) ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Freeman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Freeman, Ellen W. and Monti, Louis. Evaluation of a unique low dose intranasal aerosol for the treatment of clinically significant premenstrual symptomes NCDEU (New Clinical Drug Evaluation Unit)47th Annual Meeting,June 2007.
- See also: educational webpage about premenstrual symptoms and PMDD — http://www.acog.org/publications/patient_education/bp057.cmf